CLINICAL TRIAL: NCT04376476
Title: Host-pathogen Interactions During Paediatric and Adult SARS-CoV-2 Infection (COVID-19)
Brief Title: Host-pathogen Interactions During SARS-CoV-2 Infection
Acronym: HPI-COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL20_0342; 2020-A01102-37 (Other: ID-RCB)
Record Dates: First submitted 2020-04-28; First posted 2020-05-06 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Infection, Coronavirus; Severe Acute Respiratory Syndrome Coronavirus 2
Keywords: Severe Acute Respiratory Syndrome Coronavirus 2; COVID-19; immunology; interferon; coronavirus
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Children group E1 (Experimental): Children with confirmed asymptomatic or pauci-symptomatic COVID infection will be recruited in pediatric emergency departments, among siblings of COVID-19+ pediatric patients or through the blood collection centers set up by the occupational health services. A single visit will be scheduled at the hospital (for clinical examination, biology, immunology, virology measurements) and a phone call performed at day 14.
  Interventions: Biological: Blood sample; Biological: Low or upper respiratory tract sample; Other: phone call
- Children group E2 (Experimental): Children with confirmed COVID-19 infection requiring hospitalization will be recruited within participating centers (mostly in emergency and intensive care units). Data will be recorded (clinical examination, biology, immunology, virology measurements) during their hospital stay (day 0, day 7, in case of worsening) and a phone call performed at day 14 (or onsite visit if patient still hospitalized).
  Interventions: Biological: Blood sample; Biological: Low or upper respiratory tract sample; Biological: Stool collection or fecal swab
- Children group E3 (Experimental): Children with confirmed non-COVID-19 viral infection requiring hospitalization will be recruited within participating centers (mostly in intensive care units). At inclusion, data will be recorded (clinical examination, biology, immunology, virology measurements) and a phone call performed at day 14.
  Interventions: Biological: Blood sample; Biological: Low or upper respiratory tract sample; Biological: Stool collection or fecal swab; Other: phone call

INTERVENTIONS:
Biological: Blood sample — blood samples will be taken as below: Group E1: At day 0 Group E2: At day 0, day 7, day 14 Group E3: At day 0
Biological: Low or upper respiratory tract sample — Low or upper respiratory tract sample will be collected in order to take virology measurements:
  Group E1: At day 0 Group E2: At day 0, day 7, day 14 Group E3: At day 0
Biological: Stool collection or fecal swab — The stool collection or fecal swab will be collected in order to take virology measurements:
  Group E1: / Group E2: At day 0, day 7, day 14 Group E3: At day 0
  Arms: Children group E2; Children group E3
Other: phone call — phone calls will be performed to collect data regarding patients' symptoms at: Group E1: Day 14 Group E3: Day 14
  Arms: Children group E1; Children group E3

SUMMARY:
The new Severe acute respiratory syndrome coronavirus (SARS-CoV-2) named coronavirus disease 2019 (COVID-19) is currently responsible for a pandemic spread of febrile respiratory infections, responsible for a veritable global health crisis.

In adults, several evolutionary patterns are observed: i) a/pauci-symptomatic forms; ii) severe forms immediately linked to rare extensive viral pneumonia; and iii) forms of moderate severity, some of which progress to secondary aggravation (Day 7-Day 10). Children can be affected, but are more rarely symptomatic and severe pediatric forms are exceptional.

Like some other coronaviruses (SARS-CoV and Middle East respiratory syndrome coronavirus (MERS-CoV)), these differences in clinical expression could be based on a variability in the immunological response, notably either via inhibition of the type I interferon (IFN-I) response, or on the contrary an immunological dysregulation responsible for a "cytokine storm" associated with the aggravation. Little is known about the impact of these innate immune response abnormalities on the adaptive response. In addition, certain genetic factors predisposing to a state of "hyper-fragility" and certain viral virulence factors could also be predictive of the clinical response.

In this context, the main hypothesis is that the virological analysis and the initial biological and immunological profiles are correlated with the initial clinical presentation of COVID-19 infection. In particular, children forms and pauci-symptomatic disease in adults may be linked to a more robust innate immune response, including better production of IFN-I.

ELIGIBILITY:
Inclusion Criteria:

Group E1:

* Age from birth to <18 years old;
* Weight> 3 kilogram (kg);
* Infection with SARS-CoV-2 virus confirmed by RT-PCR on upper respiratory tract sample
* No fever or respiratory symptoms;
* Not requiring hospitalization (or hospitalization not related to a SARS-CoV-2 infection);
* Consent signed by at least one parent / holder of parental authority and assent of the child (if applicable);
* Beneficiary of a social security scheme

Group E2:

* Age from birth to <18 years old;
* Weight> 3kg;
* Infection with the SARS-CoV-2 virus confirmed by RT-PCR on a upper or low respiratory tract sample or pneumonia with scanner suggesting SARS-CoV-2 infection;
* Hospitalized in a pediatric intensive care unit or in a general pediatrics unit
* Consent signed by at least one parent / holder of parental authority and assent of the child (if applicable);
* Beneficiary of a social security scheme

Group E3:

* Age from birth to <18 years old;
* Weight> 3 kg;
* Negative SARS-CoV-2 PCR on at least one respiratory sample, and other confirmed viral infection
* Hospitalized in a pediatric intensive care unit or in a general pediatrics unit, for a respiratory reason;
* Consent signed by at least one parent / holder of parental authority and assent of the child (if applicable);
* Beneficiary of a social security scheme

Exclusion Criteria:

Group E1:

* Patients with any other inherited or acquired immune deficiency that could compromise the immunological evaluation;
* Other Suspected or proved infection
* Pregnancy.

Group E2:

* Patients with any other inherited or acquired immune deficiency that could compromise the immunological evaluation;
* Pregnancy.

Group E3:

* Patients with any other inherited or acquired immune deficiency that could compromise the immunological evaluation;
* Infection with the SARS-CoV-2 virus known among the relatives
* Pregnancy.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Initial biological profile of children with COVID-19 infection | Day 0
  Describe the immune response (biological profile in blood samples) of children and adults with COVID-19 infection and correlate it with the initial clinical presentation
  measurement of the following parameters in blood at time of inclusion: white blood cell count, C-reactive protein, procalcitonin, hepatic and renal functions, ferritin, vitamin C and D, fibrinogen, prothrombin time test and partial thromboplastin time in order to correlate them with the initial clinical presentation.
Initial immunological profile of children with COVID-19 infection | Day 0
  measurement of the following parameters in blood at time of inclusion: interferon alpha and gamma, Tumor necrosis factor (TNF) alpha, interleukins 6 and 10, transcriptomic signature of interferon, lymphocyte phenotyping and monocyte Human Leukocyte Antigen - DR isotype (HLA-DR) expression in order to correlate them with the initial clinical presentation.

SECONDARY OUTCOMES:
Clinical worsening | Within 21 days following inclusion
  Determine whether the initial biological and immunological profiles (see primary outcome measures) are predictive of a secondary worsening (i.e., admission to intensive care unit, and/or increase in NEWS-2 score, and/or increase in oxygen dependence level) of COVID-19 infection
Evolution of the immunological profile of children with COVID-19 | Within 21 days following inclusion
  measurement of the following parameters in blood at day 7, and at time of worsening: interferon alpha and gamma, TNF alpha, interleukins 6 and 10, transcriptomic signature of interferon, lymphocyte phenotyping and monocyte HLA-DR expression in order to correlate them with with the secondary worsening
Nasopharyngeal swabs SARS-CoV-2 viral loads of children with COVID-19 | Day 0
  Nasopharyngeal swabs SARS-CoV-2 viral loads (copies/mL) measured at day 0 and correlation to the initial clinical presentation
titers in specific Immunoglobulin G (IgG) antibodies of children with COVID-19 | Day 0
  Serological SARS-CoV-2 results (titers in specific Immunoglobulin G (IgG) antibodies) measured at day 0 and correlation to the initial clinical presentation
titers in specific Immunoglobulin M (IgM) antibodies of children with COVID-19 | Day 0
  Serological SARS-CoV-2 results (titers in specific Immunoglobulin M (IgM) antibodies) measured at day 0 and correlation to the initial clinical presentation
Nasopharyngeal swabs SARS-CoV-2 viral loads of children with COVID-19 | Within 21 days following inclusion
  Nasopharyngeal swabs SARS-CoV-2 viral loads (copies/mL) measured within 21 days following inclusion, and correlation to the secondary worsening
titers in specific Immunoglobulin G (IgG) antibodies of children with COVID-19 | Within 21 days following inclusion
  Serological SARS-CoV-2 results (titers in specific Immunoglobulin G (IgG) antibodies) measured within 21 days following inclusion, and correlation to the secondary worsening
titers in specific Immunoglobulin G (IgM) antibodies of children with COVID-19 | Within 21 days following inclusion
  Serological SARS-CoV-2 results (titers in specific Immunoglobulin M (IgM) antibodies) measured within 21 days following inclusion, and correlation to the secondary worsening

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Groupement Hospitalier Nord-Daupine, Bourgoin
  - Hôpital femme-mère-enfant, Bron
  - Hôpital Louis Pradel, Bron
  - Hôpital Louis Mourier, Colombes
  - Centre Hospitalier D'Annecy-Genevois, Épagny
  - Centre Hospitalo-Universitaire de Grenoble, La Tronche
  - Hopital de la Croix-Rousse, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Hôpital mère - enfant Nantes, Nantes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Nord de Saint Etienne, Saint-Priest-en-Jarez
  - Hôpital Nord-Ouest, Villefranche-sur-Saône